CLINICAL TRIAL: NCT03151200
Title: Visual Functional Connectivity and Visual Function in Amblyopia Before and After TMS and/or Binocular Treatment
Brief Title: Visual Functional Connectivity and Visual Improvement After TMS/Binocular Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated during COVID as the testing and treatment centres were closed.
Sponsor: University of Manitoba (Other)
Collaborators: University of Waterloo (Other); McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2014:117 (HS18266)
Record Dates: First submitted 2015-10-26; First posted 2017-05-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2018-10

CONDITIONS: Amblyopia
Keywords: Amblyopia treatment
MeSH Terms: conditions — Amblyopia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- binocular treatment (Active Comparator): Active treatment group will receive five days of one hour visual binocular training by playing a specifically designed falling blocks video game on a computer screen that will be individually calibrated for each person with red-green glasses with treatment effect.
  Interventions: Device: Computer based binocular treatment; Device: Transcranial magnetic stimulation
- sham treatment (Sham Comparator): Sham treatment group will receive five days of one hour sham visual binocular training by playing a specially designed falling blocks video game on a computer screen with polarized glasses with no treatment effect.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Computer based binocular treatment — Binocular amblyopia treatment involves presenting stimuli over a computer screen to the amblyopic eye those are at higher contrast compared to the stimuli that are presented to the good eye, which balances the performances of the two eyes and over time improves the amblyopic eye vision.
  Arms: binocular treatment
Device: Transcranial magnetic stimulation — TMS is a non-invasive research method that generates electrical current at the cortex that can excite neuronal activities and neuronal plasticity.
  Other Names: TMS

SUMMARY:
The purpose of this study is to assess the effectiveness of combining binocular treatment with repetitive transcranial magnetic stimulation (rTMS) in improving the vision of adults with amblyopia. This study also seeks to assess the effect of this combined treatment on cortical neural function and functional connectivity.

DETAILED DESCRIPTION:
Prior to the study, ocular misalignment and refraction abnormalities will be corrected This correction is part of standard patient care rather than a procedural component of the current study.

Procedure Participants will undergo one hour structural and functional MRI prior to their treatment. We will perform an interim analysis of the fMRI results once five amblyopic patients have completed the fMRI study. If the data shows significant differences in the resting state visual network in amblyopia patients compared to the existing normal visual resting state, we will pursue the fMRI study with the remaining 15 participants. Misalignment of the eyes will be corrected prior to a patients' participation by using prisms (if medically indicated). This correction is part of standard patient care rather than a procedural component of the current study. Participants will be randomly appointed to initially be in either the sham or the treatment group (10 patients in each group). All patients will receive five days of one hour visual binocular training by playing a specially designed falling blocks videogame on a computer screen that will be individually calibrated for each person. Group one will receive 18 minutes of rTMS at the beginning of their visual training every day for 5 days. Group two will receive 18 minutes of TMS followed by sham visual training every day for 5 days. At the end of five days, participants will switch groups. Participants will be blind as to whether they receive sham or real binocular treatment on each occasion.

A sensorimotor visual profile, including visual acuity, suppression, stereovision, binocularity, contrast sensitivity and eye alignment, will be completed for each patient at baseline, after five sessions, and at the end of the treatment. This profile will be completed using the PVVAT system, Worth-4-Dot test, Randot stereovision test, anaglyphic dichoptic coherence motion threshold with red-green glasses (using Psykinematix vision system), cross cover test with prism bars. fMRI will be repeated post-treatment only for individuals who showed abnormal fMRI at baseline. This second scan will investigate whether the treatment affected and normalized the resting state visual network.

Functional MRI:

All scanning will be performed on a 3.0 T Siemens Tim Trio scanner equipped with a 12-channel head coil. Scanning will take place on up to three visits: Pre-treatment (retinotopic mapping), and two post treatment scans.

Pre-treatment: structural, resting state and BOLD functional MRI (fMRI) data will be acquired. Participants will complete a structural MRI scan at the beginning of each MRI session. This is a high-resolution 3-dimensional image of the whole brain (Imaging parameters: MPRAGE, 1mm thick slices, zero spacing between slices, TR = 1900 ms, TE = 2.2 ms, in plane resolution of 0.94 x 0.94, 256 x 256 matrix size with a 24 cm field of view, 176 volumes, resulting in a 8 minute 6 second scan time.

After the high-resolution image has been acquired, the resting state functional MRI data will be acquired with the following parameters: Siemens echo planar imaging (EPI) sequence, 3 mm thick slices, zero spacing between slices, repetition time of 3000 ms, echo time of 30 ms, flip angle of 90°, 64 x 64 matrix size, 24 cm field of view, 140 volumes, resulting in a 7 minute 9 second scan time. During this session the patients will close their eyes and rest.

Following the resting state fMRI session we will perform task-based and retinotopic mapping using standard wedge and ring protocols to evoke blood oxygen level-depended (BOLD) response in the visual cortex. (Li X, Dumoulin SO, Mansouri B, Hess RF. The fidelity of the cortical retinotopic map in human amblyopia. Eur J Neurosci. 2007;25:1265-1277.29). Functional data will be acquired using a T2-weighted gradient echo EPI sequence (retinotopic mapping, TR = 1200 ms, TE = 30 ms, flip angle = 65°, voxel resolution 2.5 x 2.5 x 2.5 mm; post treatment scans, TR = 2000 ms, TE = 30 ms, flip angle = 90°, voxel resolution = 3.0 x 3.0 x 3.0 mm). Stimuli will be presented monocularly and each eye will be mapped separately. Borders of retinotopic areas and corresponding regions of interest will be defined using an averaged map of the left and right eye in each participant. During fMRI, participants will be presented with visual stimuli (viewed over an MRI compatible white screen through a coil-mounted mirror) and perform a reaction time task where they will simply press a button when they detect a change in the fixation point. The task will be unrelated to the stimuli used.

The subsequent fMRI scanning sessions will be performed after two week of Transcranial Magnetic stimulation (TMS) and binocular treatment, which will assess the effect of rTMS plus sham/real binocular treatment on the response of the visual cortex to inputs from the amblyopic versus fellow fixing eye. We will use the localizing information from the first session. The resting state and task-based fMRI will be repeated.

1. Pre -treatment visit:

a. Localizer to find slice plan (1-2 min) b. MPRAGE anatomical (7-10 min) c. Resting state - eyes closed stay awake (7-10 min) d. Retinotopic mapping (48 min PLUS time to alternate eye patch between runs) i. 4 scans of block design amblyopic eye covered

1. 2 eccentricity,
2. 2 polar angle,
3. 2 clockwise,
4. 2 counterclockwise, ii. 4 scans of block design fellow fixing eye covered

One week of either Group A) rTMS and true binocular treatment or Group B) rTMS and sham binocular treatment 2. Post treatment visit:

1. Localizer (1-2 min)
2. MPRAGE anatomical (7-10 min)
3. Resting state - eyes closed stay awake (
4. not retinotopic mapping
5. fMRI block design

i. checkerboard stimulus 4 scans per session per eye One week of CROSS OVER treatment Group A) rTMS and sham binocular treatment or Group B) rTMS and binocular treatment fMRI analysis Resting state fMRI data will be pre-processed to reduce artifacts and noise-related signal components. Following pre-processing, data will be analyzed at the individual level using Independent Component Analysis. The individually analyzed data will then be standardized to stereotactic space using a Talairach atlas. The standardized data will be run through a Self-Organized Grouped ICA which will summarize the ICA data from all participants. An analysis of variance will be used to assess differences in functional connectivity in brain regions between the groups (pre- and post-rTMS treatment).

Potential harms and benefits It is our hope that as a result of their participation in this study, patients will see an improvement in many aspects of their vision, including overall visual acuity and contrast sensitivity.

There is a chance that improving vision in the weak eye may result in double vision if the position of the eyes (alignment) is suboptimal. This double vision may spontaneously subside over time as the training effect wears off (in the absence of further training). If double vision persists, participants may have to be referred to neurology, optometry or ophthalmology clinics for symptom management. Patching over the weak eye may be required in order to eliminate the double vision, decreasing vision in the weak eye in an effort to returning vision to what it was before participation in the study. Other treatments for double vision include optical correction with glasses that contain prisms or surgical intervention to align the two eyes. The latter methods help fuse images from the two eyes in most of cases.

The rTMS procedures proposed for this study are well within recommended safety guidelines, so the risk of adverse events is slim. TMS can cause twitching of the scalp or face muscles during stimulation, which may be uncomfortable. About 1 out of 10 subjects report a headache after the TMS measurement, which is usually mild and transient. If needed, the headache can be treated with mild over-the-counter pain medicine, such as acetaminophen/Tylenol. The risk of seizure from rTMS is elevated in individuals with a history of epilepsy or a family history of seizures, which is why these conditions are exclusion criteria for this study.

ELIGIBILITY:
Inclusion Criteria:

* A total of 20 strabismic or mixed amblyopic adult patients (eighteen or older) will be recruited from Dr. Mansouri's practice. Patients will be asked for their permission to be contacted by a research assistant with regard to the study. A research assistant will then contact patients and inform them about the study, its procedures, and its voluntary nature. Patients will not be contacted without their previous permission.

Exclusion Criteria:

* Given the use of rTMS and MRI in this study, participants will be excluded if they have any contraindications to these procedures. Contraindications include: the presence of metal clips or implants in the body (such as pacemakers, defibrillators or neural stimulators), metallic dental work, severe claustrophobia, epilepsy, a family history of seizures, or the taking of epileptogenic medications. Pregnant individuals will also be excluded as a precaution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Improvement of visual acuity in amblyopic eyes after TMS/binocular treatment | 2 weeks treatment

SECONDARY OUTCOMES:
Improvement of stereovision and reduction in suppression in amblyopic patients after TMS/binocular treatment | 2 weeks treatment

OTHER OUTCOMES:
Brain function and connectivity changes after TMS/binocular treatment | 2 weeks treatment

CONTACTS AND LOCATIONS:
Locations (1):
- VGH Adult Medical Clinic, Winnipeg, Manitoba, Canada